CLINICAL TRIAL: NCT07184957
Title: Prospective Database of Clinical Outcomes Following Cryotherapy for Ablation of Clinically Localized Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 17-00354
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men with Prostate Cancer: Men who receive cryotherapy for ablation of clinically localized prostate cancer.

SUMMARY:
This will be a prospectively maintained research database. The purpose is to record baseline parameters and treatment outcomes following of Cryotherapy for ablation of clinically localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of focal prostate cancer confined to the prostate based on MRI imaging and prostate biopsy
* Patients with clinically localized prostate cancer (no evidence for or concern for metastatic spread of cancer outside of the prostate) will be counseled regarding treatment options. Those selecting focal Cryo prostate ablation will then be offered inclusion into this data collection.

Exclusion Criteria:

* Men that are not diagnosed with prostate cancer.
* Men that are diagnosed with clinically localized prostate cancer, but select other treatment options as their desired treatment.

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who receive cryotherapy for ablation of clinically localized prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Complications | Up to Year 15
PSA-Progression Free Survival | Up to Year 15
  Length of time following cryotherapy for ablation treatment of prostate cancer that a patient lives without their prostate-specific antigen (PSA) levels rising significantly enough to indicate disease recurrence, or without dying from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: James Wysock, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: James.Wysock@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to James.Wysock@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.